CLINICAL TRIAL: NCT00957073
Title: Health Outcomes Prospective Evaluation for Heart Failure With Ejection Fraction (EF) ≥ 40%
Brief Title: Rheos System for the Treatment of HFpEF Heart Failure
Acronym: HOPE4HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CVRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 360017-001
Record Dates: First submitted 2009-08-10; First posted 2009-08-12 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Heart Failure
Keywords: Heart Failure; Diastolic dysfunction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Device (Experimental): Rheos® system
  Interventions: Device: Rheos® system
- Medical Management (No Intervention): Medical Management Therapy

INTERVENTIONS:
Device: Rheos® system — Implant procedure
  Other Names: Rheos® Baroreflex Activation Therapy®; Neo Legacy® System; BAROSTIM NEO® LEGACY System
  Arms: Device

SUMMARY:
The purpose of this clinical investigation (NCT00957073) is to continue long-term follow-up of device arm subjects enrolled in the HOPE4HF Trial, utilizing the BAROSTIM NEO™ LEGACY device for Implantable Pulse Generator (IPG) replacements.

DETAILED DESCRIPTION:
The initial trial design randomized subjects in a 2:1 ratio to receive a Rheos system plus medical management (Device Arm) or to receive medical management alone (Medical Management Arm). On March 24, 2011, the study closed to enrollment before adequate endpoint data was collected and before enrollment was completed; 19 subjects had been randomized, 10 device and 9 medical management. Medical management subjects were withdrawn from the study and subjects who had been implanted with the device were given the opportunity to continue in the study under long-term follow-up; 8 of the 10 device subjects continued in the study. Long-term follow-up visits occurred at 15 and 18 months post-randomization; visits occur semi-annually until study closure.

The study was not stopped for safety or futility, but for business/strategic reasons due to production of a new generation of the device.

ELIGIBILITY:
Inclusion Criteria:

1. Currently implanted with the Rheos device and actively participating in the HOPE4HF Trial (G090001).
2. Have signed a CVRx, FDA and Institutional Review Board (IRB) approved informed consent form for participation in this study.

Exclusion Criteria:

1. Treating physician decision that the subject should not continue with therapy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-08; Primary Completion 2012-10 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
To ascertain long-term adverse events for subjects implanted with the device. | Trial duration
  To systematically and actively ascertain the type, frequency, severity and timing of long-term adverse events in subjects implanted with the device.

CONTACTS AND LOCATIONS:
Overall Officials: William Abraham, MD, Principal Investigator — Ohio State University; Fred Weaver, MD, Principal Investigator — University of Southern California; Michael Zile, MD, Study Chair — Medical University of South Carolina; Faiez Zannad, MD, Principal Investigator — Inserm Centre d'Investigation, CHU de Nancy; JoAnn Lindenfield, MD, Principal Investigator — Vanderbilt Heart and Vascular Institute
Locations (22):
- United States (22):
  - Cardiology Associates of Mobile, Inc., Mobile, Alabama
  - Apex Cardiology Consultants, Inglewood, California
  - University of Southern California, Los Angeles, California
  - St. Francis Hospital and Medical Center, Hartford, Connecticut
  - Florida Hospital Cardiovascular Institute/Florida Heart Group, Orlando, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Heart and Vascular Institute of Florida, St. Petersburg, Florida
  - Florida Cardiovascular Institute, Tampa, Florida
  - The Care Group, Indianapolis, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Liberty Cardiovascular Specialists, Liberty, Missouri
  - Washington University, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - Forsyth Cardiovascular Research, Winston-Salem, North Carolina
  - Lindner Research Center, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Northwest Ohio Cardiology Consultants, Toledo, Ohio
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - Drexel University, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- [Derived] Georgakopoulos D, Little WC, Abraham WT, Weaver FA, Zile MR. Chronic baroreflex activation: a potential therapeutic approach to heart failure with preserved ejection fraction. J Card Fail. 2011 Feb;17(2):167-78. doi: 10.1016/j.cardfail.2010.09.004. Epub 2010 Oct 29. PMID 21300307